CLINICAL TRIAL: NCT04442074
Title: Characteristics in Doppler Ultrasound of the Carotid Diaphragm Responsible for an Ischemic Stroke
Acronym: DIADOP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: DIADOP
Record Dates: First submitted 2020-06-17; First posted 2020-06-22 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke Patients: These patients were hospitalized in the neurology / neurovascular department of the Paris Saint-Joseph Hospital Group, for the management of a transient ischemic infarction or accident for which the diagnosis of ipsilateral carotid diaphragm was accepted, between April 2017 and April 2020.

SUMMARY:
Carotid diaphragms are a non-atheromatous arterial cause of cerebral infarction, especially in young people (≤65 years old). This anomaly is more common in the African or African-American population, although it is more and more often discovered in young Caucasians. This cause of cerebrovascular accident (CVA), known until the 1970s, was later forgotten until a recent revival of interest, probably in connection with the improvement of imagery but also by the discovery that these lesions have a high rate of recurrence in the absence of interventional care. In a Brazilian study, the carotid diaphragm was reported in 10% of patients under the age of 60.

The carotid diaphragm is a non-atheromatous overgrowth of the intima of the arterial wall. It appears in imagery in the form of an endoluminal web wider than it is tall. Its preferred seat is the carotid bulb. It is a source, by an embologenic mechanism, of cerebral infarction starting from local thrombus developed within large cerebral arteries. In histology, the lesions are different from atherosclerosis and characterized by a thickening of the intima with proliferation of loose and strewed spindle cells mainly involving the intima.

An atheromatous plaque or dissection with detachment of the intima are the two main differential diagnoses of the carotid web. However, the appearance of a diaphragm implanted on a regular wall and the absence of any other localization of atheroma distinguish the lesion of the carotid web from that of a focal atheromatous plate. In addition, the very proximal localization of the carotid web, from the emergence of the internal carotid artery, does not suggest a dissection, the localization of which is usually downstream of the bulb.

The baseline exam to detect a carotid diaphragm is a carotid angiography scan, but the abnormalities are often inconspicuous, making diagnosis difficult. We can be led in case of doubt to perform a conventional arteriography, which remains the "gold standard". The latter, dynamic examination compared to the CT scan, shows above all a stasis of blood flow in the recess created by the diaphragm, stasis at the origin of the formation of thrombi. It has been suspected that the maximum risk of infarction is upon waking, at the time of verticalization, with mobilization of the thrombus.

Therapeutically, the discovery of a symptomatic carotid diaphragm (ischemic swallowing accident) justifies radical treatment. The risk of recurrence of a patient on antithrombotic (antiplatelet or anticoagulant) being too high, it is proposed either surgery, or carotid angioplasty with stent placement. No comparative study of the 2 techniques has been carried out.

Besides radiological examinations, ultrasound is another technique for studying the cervical arteries. It is reputed to be of little contribution in the search for a carotid diaphragm, but few publications exist to date even though the cervical Doppler is often the first arterial examination carried out after an ischemic stroke. Two series reported Doppler ultrasound data in the carotid diaphragm. A recent retrospective study evaluated, in multimodal imaging [Doppler, CT scan of the Supra-Aortic Trunks (ASD) and conventional arteriography], 30 patients (60 carotids) with diaphragm or atherosclerosis. The correlation between conventional arteriography and CT angiography was perfect, but the correlation between Doppler and CT angiography for diaphragm diagnosis was moderate. In another series studying 15 diaphragms diagnosed by CT angiography, the retrospective analysis of doppler reports revealed that 40% were considered normal and 60% mentioned nonspecific hyperechoic lesions, but this work remained in the form of a presentation. at a congress. With the improvement of the technique and the resolution of the Doppler ultrasound as well as the knowledge of the particular ultrasound characteristics, it seems to us that this examination could regain a place in the diagnosis of the pathology. The carotid diaphragm is also largely unknown to vascular doctors practicing cervical Doppler ultrasound.

This descriptive study of the diagnostic contribution of the echo-doppler for a carotid diaphragm has for perspective the establishment of a prospective study of the contribution of a combined expertise angiologist-neurologist in the echo-Doppler for patients <60 years hospitalized for an ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is> 18 years old and ≤65 years old
* Patients treated in the neurology department for an infarction or transient ischemic attack for which the diagnosis of ipsilateral carotid diaphragm was accepted, between April 2017 and April 2020
* French speaking patients

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient objecting to the use of his data for this research

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were hospitalized in the neurology / neurovascular department of the Paris Saint-Joseph Hospital Group, for the management of a transient ischemic infarction or accident for which the diagnosis of ipsilateral carotid diaphragm was accepted, between April 2017 and April 2020.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2020-06-13 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Doppler ultrasound sensitivity for the carotid diaphragm | Day 1
  This outcome corresponds to the number of echo-doppler reports for which the diagnosis of carotid diaphragm is mentioned, correlated to the number of echo-doppler images presenting anomalies suggestive of carotid diaphragm.

SECONDARY OUTCOMES:
Description of Anomalies suggestive of carotid diaphragm on Doppler ultrasound | Day 1
  This outcome corresponds to the description of the evocative anomalies visualized in echo-dopple (visualization of an intimal spur, of an associated thrombus, of a morphological / hemodynamic stenosis, of turbulence of the flow).
Sensitivity of the Doppler ultrasound with that of the reference vascular examinations | Day 1
  This outcome corresponds to to the comparison of the number of patients with a diagnosis of carotid diaphragm according to the examination carried out using the review of the additional imagery carried out and the anatomopathological result when this was carried out.

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Tamazyan, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Result] Haussen DC, Grossberg JA, Bouslama M, Pradilla G, Belagaje S, Bianchi N, Allen JW, Frankel M, Nogueira RG. Carotid Web (Intimal Fibromuscular Dysplasia) Has High Stroke Recurrence Risk and Is Amenable to Stenting. Stroke. 2017 Nov;48(11):3134-3137. doi: 10.1161/STROKEAHA.117.019020. Epub 2017 Oct 10. PMID 29018133
- [Result] Coutinho JM, Derkatch S, Potvin AR, Tomlinson G, Casaubon LK, Silver FL, Mandell DM. Carotid artery web and ischemic stroke: A case-control study. Neurology. 2017 Jan 3;88(1):65-69. doi: 10.1212/WNL.0000000000003464. Epub 2016 Nov 18. PMID 27864523
- [Result] Madaelil TP, Grossberg JA, Nogueira RG, Anderson A, Barreira C, Frankel M, Haussen DC. Multimodality Imaging in Carotid Web. Front Neurol. 2019 Mar 12;10:220. doi: 10.3389/fneur.2019.00220. eCollection 2019. PMID 30915028